CLINICAL TRIAL: NCT04499534
Title: Influenza Vaccine Study in BRCA1 or BRCA2 Carriers
Brief Title: BRCA1/2 Flu Vaccine
Status: Active, not recruiting | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 11119; 834194 (Other: University of Pennsylvania Protocol Number)
Record Dates: First submitted 2020-06-16; First posted 2020-08-05 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: BRCA1 Mutation; BRCA2 Mutation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: Seasonal influenza vaccine — To evaluate immune function in BRCA1/2 mutation carriers without cancer following seasonal influenza vaccination

SUMMARY:
To evaluate immune function in BRCA1/2 mutation carriers without cancer, specifically to determine whether immune function in healthy individuals with germline loss of function BRCA1/2 mutations, impacts overall immune health and fitness.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Over age 25
* BRCA1 or BRCA2 pathogenic or likely pathogenic mutation
* No personal cancer history apart from non melanoma skin cancer, localized thyroid cancer, in situ cancers of any type
* Participants must sign the informed consent form

Exclusion Criteria:

* Are allergic to influenza vaccination
* Have received influenza vaccination within the past 6 months
* Require prednisone, methotrexate, or other immunosuppressing medications
* Have HIV infection
* Have a history of solid organ tumor or bone marrow transplant
* Require combination immunotherapy;
* Are on other studies requiring blood draws that might exceed 450 mL total during the period of the influenza vaccine study

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients 25 years and older, seen at Cancer Risk Evaluation Program (CREP) in the Perelman Center for Advanced Medicine with BRCA1 or BRCA2 mutation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-10-28 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
To evaluate immune function in female BRCA1/2 mutation carriers without cancer following seasonal influenza vaccination | 2 years
  Analysis of the primary objective will depend on determination of the strain-specific neutralizing antibody titer change from day 0 to the last study visit, performed as the standard assay as described by the World Health Organization (WHO).

SECONDARY OUTCOMES:
Exploratory analysis- phenotypic evaluation of B cell | 2 years
  Phenotypic evaluation of B and T cell responses to vaccine at each timepoint. Phenotypic analysis involves flow cytometry on peripheral blood mononuclear cells (PBMC) from all subjects (10 mL blood per subject).
Exploratory analysis - transcriptional evaluation | 2 years
  Transcriptional evaluation of B and T cell responses to vaccine on day 7-10 timepoint. Transcriptional analyses including quantitative real-time PCR (RT-qPCR) and RNA sequencing (RNAseq) may be performed on a subset of the study subjects on the day 7-10 time point.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Domchek, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mouw KW, Goldberg MS, Konstantinopoulos PA, D'Andrea AD. DNA Damage and Repair Biomarkers of Immunotherapy Response. Cancer Discov. 2017 Jul;7(7):675-693. doi: 10.1158/2159-8290.CD-17-0226. Epub 2017 Jun 19. PMID 28630051
- [Background] Brodin P, Jojic V, Gao T, Bhattacharya S, Angel CJ, Furman D, Shen-Orr S, Dekker CL, Swan GE, Butte AJ, Maecker HT, Davis MM. Variation in the human immune system is largely driven by non-heritable influences. Cell. 2015 Jan 15;160(1-2):37-47. doi: 10.1016/j.cell.2014.12.020. PMID 25594173
- [Background] Casanova JL, Abel L, Quintana-Murci L. Immunology taught by human genetics. Cold Spring Harb Symp Quant Biol. 2013;78:157-72. doi: 10.1101/sqb.2013.78.019968. Epub 2013 Oct 3. PMID 24092470
- [Background] Lucas CL, Lenardo MJ. Identifying genetic determinants of autoimmunity and immune dysregulation. Curr Opin Immunol. 2015 Dec;37:28-33. doi: 10.1016/j.coi.2015.09.001. Epub 2015 Oct 2. PMID 26433354
- [Background] Mak TW, Hakem A, McPherson JP, Shehabeldin A, Zablocki E, Migon E, Duncan GS, Bouchard D, Wakeham A, Cheung A, Karaskova J, Sarosi I, Squire J, Marth J, Hakem R. Brca1 required for T cell lineage development but not TCR loci rearrangement. Nat Immunol. 2000 Jul;1(1):77-82. doi: 10.1038/76950. PMID 10881179
- [Background] Cheung AM, Hande MP, Jalali F, Tsao MS, Skinnider B, Hirao A, McPherson JP, Karaskova J, Suzuki A, Wakeham A, You-Ten A, Elia A, Squire J, Bristow R, Hakem R, Mak TW. Loss of Brca2 and p53 synergistically promotes genomic instability and deregulation of T-cell apoptosis. Cancer Res. 2002 Nov 1;62(21):6194-204. PMID 12414647
- [Background] Centers for Disease Control and Prevention (CDC). Estimates of deaths associated with seasonal influenza --- United States, 1976-2007. MMWR Morb Mortal Wkly Rep. 2010 Aug 27;59(33):1057-62. PMID 20798667
- [Background] Herati RS, Reuter MA, Dolfi DV, Mansfield KD, Aung H, Badwan OZ, Kurupati RK, Kannan S, Ertl H, Schmader KE, Betts MR, Canaday DH, Wherry EJ. Circulating CXCR5+PD-1+ response predicts influenza vaccine antibody responses in young adults but not elderly adults. J Immunol. 2014 Oct 1;193(7):3528-37. doi: 10.4049/jimmunol.1302503. Epub 2014 Aug 29. PMID 25172499
- [Background] Schaerli P, Willimann K, Lang AB, Lipp M, Loetscher P, Moser B. CXC chemokine receptor 5 expression defines follicular homing T cells with B cell helper function. J Exp Med. 2000 Dec 4;192(11):1553-62. doi: 10.1084/jem.192.11.1553. PMID 11104798